CLINICAL TRIAL: NCT03298867
Title: A Phase 3, Randomized, Double-Masked, Placebo-Controlled, Parallel-Group, Multicenter Study Evaluating Teprotumumab (HZN-001) Treatment in Subjects With Active Thyroid Eye Disease
Brief Title: Treatment of Graves' Orbitopathy (Thyroid Eye Disease) to Reduce Proptosis With Teprotumumab Infusions in a Randomized, Placebo-Controlled, Clinical Study
Acronym: OPTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZNP-TEP-301; 2017-002763-18 (EudraCT Number)
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Results first posted 2020-03-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Thyroid Eye Disease; Graves' Orbitopathy
Keywords: Proptosis; Human monoclonal antibody; insulin-like growth factor-1 receptor; Thyroid-Associated Ophthalmopathy; Autoimmune Thyroid Disease; Graves' Orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy; Exophthalmos | interventions — teprotumumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teprotumumab 20 mg/kg (Active Comparator): Approximately 38 participants will receive 8 infusions of teprotumumab q3W for a total of 21 weeks. Teprotumumab 10 mg/kg will be administered on Day 1 and teprotumumab 20 mg/kg will be administered q3W for the remaining 7 infusions.
  Interventions: Biological: Teprotumumab
- Placebo (Placebo Comparator): Approximately 38 participants will receive 8 infusions of placebo q3W for a total of 21 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Teprotumumab — Teprotumumab is a fully human anti-IGF-1R mAb. Teprotumumab will be provided in single-dose 20 mL glass vials as a freeze-dried powder. Each vial of teprotumumab must be reconstituted with 10 mL of water for injection. Reconstituted teprotumumab solution must be further diluted in 0.9% (w/v) sodium chloride (NaCl) solution prior to administration. Teprotumumab will be administered in 100 mL or 250 mL infusion bags (100 mL infusion bags for doses up to 1800 mg and 250 mL infusion bags for doses > 1800 mg).
  Other Names: HZN-001
  Arms: Teprotumumab 20 mg/kg
Other: Placebo — Placebo will consist of normal saline (0.9% NaCl) solution and will be administered in 100 mL or 250 mL infusion bags, as would be appropriate, per weight-based dosing volumes (100 mL infusion bags for doses up to 1800 mg and 250 mL infusion bags for doses > 1800 mg).
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The overall objective is to investigate the efficacy, tolerability, and safety of teprotumumab (a fully human monoclonal antibody [mAb] inhibitor of the insulin-like growth factor-1 receptor [IGF-1R]) administered once every 3 weeks (q3W) for 21 weeks with a final assessment at Week 24, in comparison to placebo, in the treatment of participants with moderate-to-severe active thyroid eye disease (TED).

DETAILED DESCRIPTION:
This is a randomized, double-masked, placebo-controlled, parallel-group, multicenter study. Approximately 76 participants (38/group) who meet the study eligibility criteria will be randomized on Day 1 in a 1:1 ratio (stratified by tobacco use status) to receive 8 infusions of teprotumumab or placebo q3W. All participants will enter a 24-week double-masked Treatment Period, during which study drug will be infused on Day 1 (Baseline), and Weeks 3, 6, 9, 12, 15, 18, and 21 (with a final visit at Week 24). All study drug dosing will be performed at the clinic under the supervision of clinic staff. On each dosing day, scheduled assessments (except for adverse event [AE] and concomitant medication use monitoring, which will be monitored throughout the clinic visit) will be completed prior to study drug dosing.

At the end of the double-masked Treatment Period (Week 24), participants who are proptosis non-responders (study eye has < 2 mm decrease in proptosis) will be eligible to enter an open-label extension study in which participants receive 8 infusions of teprotumumab in an open-label fashion.

At Week 24, proptosis responders, as well as non-responders who choose not to enroll in the open-label extension study, will enter a 48-week Follow-Up Period, during which study drug will not be administered and clinic visits are scheduled for Weeks 28, 36, 48, 60, and 72. Participants who are considered responders at Week 24 but who meet criteria for re-treatment due to relapse during the Follow-Up Period may enroll in the open-label extension study.

Participants who complete the Week 72 Visit will be contacted 6 and 12 months later via phone or email by research staff to enquire if any treatment for TED has been received since last study contact.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female participant between the ages of 18 and 80 years, inclusive, at Screening.
3. Clinical diagnosis of Graves' disease associated with active TED with a Clinical Activity Score (CAS) ≥ 4 (on the 7-item scale) for the most severely affected eye at Screening and Baseline.
4. Moderate-to-severe active TED (not sight-threatening but has an appreciable impact on daily life), usually associated with one or more of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, exophthalmos ≥ 3 mm above normal for race and gender, and/or inconstant or constant diplopia.
5. Onset of active TED symptoms (as determined by participant records) within 9 months prior to Baseline.
6. Participants must be euthyroid with the baseline disease under control or have mild hypo- or hyperthyroidism (defined as free thyroxine [FT4] and free triiodothyronine [FT3] levels < 50% above or below the normal limits) at Screening. Every effort should be made to correct the mild hypo- or hyperthyroidism promptly and to maintain the euthyroid state for the full duration of the clinical trial.
7. Does not require immediate surgical ophthalmological intervention and is not planning corrective surgery/irradiation during the course of the study.
8. Alanine aminotransferase (ALT) or AST ≤ 3 times the upper limit of normal (ULN) or serum creatine <1.5 times the ULN according to age at Screening.
9. Diabetic participants must have well-controlled stable disease (defined as HbA1C < 9.0% with no new diabetic medication [oral or insulin] or more than a 10% change in the dose of a currently prescribed diabetic medication within 60 days prior to Screening).
10. Women of childbearing potential (including those with an onset of menopause <2 years prior to Screening, non-therapy-induced amenorrhea for <12 months prior to Screening, or not surgically sterile [absence of ovaries and/or uterus]) must have a negative serum pregnancy test at Screening and negative urine pregnancy tests at all protocol-specified timepoints (i.e., prior to each dose and through Week 48 of the Follow-Up Period); participants who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the trial, one of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started at least one full cycle prior to Baseline and continue for 180 days after the last dose of study drug. Highly effective contraceptive methods (with a failure rate less than 1% per year) when used consistently and correctly, includes implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence or vasectomized partner.
11. Male participants must be surgically sterile or, if sexually active with a female partner of childbearing potential, must agree to use barrier contraceptive method from Screening through 180 days after the last dose of study drug.
12. Participant is willing and able to comply with the study protocol and evaluations for the duration of the study.

Exclusion Criteria:

1. Decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months.
2. Corneal decompensation unresponsive to medical management.
3. Decrease in CAS of ≥ 2 points in the study eye between Screening and Baseline.
4. Decrease in proptosis of ≥ 2 mm in the study eye between Screening and Baseline.
5. Previous orbital irradiation or surgery for TED.
6. Any steroid use (intravenous [IV] or oral) with a cumulative dose equivalent to ≥ 1 g of methylprednisolone for the treatment of TED. Previous steroid use (IV or oral) with a cumulative dose of <1 g methylprednisolone or equivalent for the treatment of TED and previous use of steroid eye drops is allowed if the corticosteroid was discontinued at least 4 weeks prior to Screening.
7. Corticosteroid use for conditions other than TED within 4 weeks prior to Screening (topical steroids for dermatological conditions and inhaled steroids are allowed).
8. Selenium and biotin must be discontinued 3 weeks prior to Screening and must not be restarted during the clinical trial; however, taking a multivitamin that includes selenium and/or biotin is allowed.
9. Any previous treatment with rituximab or tocilizumab. Use of any other non-steroid immunosuppressive agent within 3 months prior to Screening.
10. Use of an investigational agent for any condition within 60 days prior to Screening or anticipated use during the course of the trial.
11. Identified pre-existing ophthalmic disease that, in the judgment of the Investigator, would preclude study participation or complicate interpretation of study results.
12. Bleeding diathesis that in the judgment of the Investigator would preclude inclusion in the clinical trial.
13. Malignant condition in the past 12 months (except successfully treated basal/squamous cell carcinoma of the skin).
14. Pregnant or lactating women.
15. Current drug or alcohol abuse, or history of either within the previous 2 years, in the opinion of the Investigator or as reported by the participant.
16. Biopsy-proven or clinically suspected inflammatory bowel disease.
17. Known hypersensitivity to any of the components of teprotumumab or prior hypersensitivity reactions to mAbs.
18. Any other condition that, in the opinion of the Investigator, would preclude inclusion in the study.
19. Previous enrollment in this study or participation in a prior teprotumumab clinical trial.
20. Human immunodeficiency virus (HIV), hepatitis C or hepatitis B infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (9):
  - Macro, Llc, Beverly Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Lennar Foundation Medical, Coral Gables, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Kellogg Eye Center at University of Michigan, Ann Arbor, Michigan
  - Casey Eye Institute at Oregon Health and Science University, Portland, Oregon
  - Hamilton Eye Institute at University of Tennessee Health Science Center, Memphis, Tennessee
  - Eye Wellness Center, Houston, Texas
  - Medical College of Wisconsin, The Eye Institute, Milwaukee, Wisconsin
- Germany (2):
  - University Hospital Essen, Department of Ophthalmology, Essen
  - Johannes Gutenberg University Medical Center, Mainz
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - University of Pisa, Department of Clinical and Experimental Medicine, Pisa
  - University of Pisa,Department of Clinical and Experimental Medicine, Endocrinology Unit, Pisa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Result] Douglas RS, Kahaly GJ, Patel A, Sile S, Thompson EHZ, Perdok R, Fleming JC, Fowler BT, Marcocci C, Marino M, Antonelli A, Dailey R, Harris GJ, Eckstein A, Schiffman J, Tang R, Nelson C, Salvi M, Wester S, Sherman JW, Vescio T, Holt RJ, Smith TJ. Teprotumumab for the Treatment of Active Thyroid Eye Disease. N Engl J Med. 2020 Jan 23;382(4):341-352. doi: 10.1056/NEJMoa1910434. PMID 31971679
- [Derived] Jain AP, Gellada N, Ugradar S, Kumar A, Kahaly G, Douglas R. Teprotumumab reduces extraocular muscle and orbital fat volume in thyroid eye disease. Br J Ophthalmol. 2022 Feb;106(2):165-171. doi: 10.1136/bjophthalmol-2020-317806. Epub 2020 Nov 10. PMID 33172865
- See also: Related Info — https://www.tepezza.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Eight infusions of placebo every 3 weeks (q3W) for a total of 21 weeks.
- Teprotumumab 20 mg/kg: Eight infusions of teprotumumab every q3W for a total of 21 weeks. Teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
Period: Double-Masked 24-Week Treatment Period
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Started | 42 | 41
Completed | 40 (36 participants who completed the double-masked treatment period as nonresponders chose to enroll in the OPTIC-X open-label extension study (NCT03461211).) | 39 (3 participants who completed the double-masked treatment period as nonresponders chose to enroll in the OPTIC-X open-label extension study (NCT03461211).)
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: 48-Week Follow-Up Period (Weeks 24-72)
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Started | 4 | 36
Completed | 3 | 20
Not Completed | 1 | 16
Not completed — Relapsed/Entered OPTIC-X | 1 | 9
Not completed — Relapsed/Did not enter OPTIC-X | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other, Not Specified | 0 | 1
Not completed — Mis-classified as Responders | 0 | 2
Period: 48-Week Follow-Up Contact (Weeks 96-120)
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Started | 3 | 20
Completed | 3 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eight infusions of placebo q3W for a total of 21 weeks.
- Teprotumumab 20 mg/kg: Eight infusions of teprotumumab q3W for a total of 21 weeks. Teprotumumab 10 mg/kg administered on Day 1 and teprotumumab 20 mg/kg administered q3W for the remaining 7 infusions.
- Total: Total of all reporting groups
Arm/Group | Placebo | Teprotumumab 20 mg/kg | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.96) | 51.6 (12.63) | 50.2 (12.79)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 38 | 32 | 70
  ≥65 years | 4 | 9 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 41 | 39 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3
  Black or African American | 2 | 4 | 6
  White | 37 | 35 | 72
  More Than 1 Race | 2 | 0 | 2
Tobacco use status - as randomized [Count of Participants; unit: Participants]
  Non-User | 33 | 32 | 65
  User | 9 | 9 | 18
Tobacco use status - actual [Count of Participants; unit: Participants] — Actual tobacco use status reflects the status as reported on the substance use case report form. One participant was randomized in error to the tobacco user stratum as this subject was reported as a non-user (former tobacco use status) on the substance use case report form.
  Participants
    Non-User | 34 | 32 | 66
    User | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Proptosis Responders at Week 24
Description: Proptosis responders were defined as participants with a ≥2 mm reduction from Baseline in proptosis in the study eye, without deterioration (≥2 mm increase) of proptosis in the fellow eye at Week 24.
Time Frame: Week 24
Population: Intent-to-treat population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Number analyzed (Participants) | 42 | 41
percentage of participants | 9.5 | 82.9
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab 20 mg/kg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Two-sided p-value calculated assuming the test statistic was distributed as a standard normal random variable; Stratified difference in percentages = 73.45, 95% CI 2-sided [58.89 to 88.01], Standard Error of Mean 7.43 — Stratified difference (teprotumumab - placebo) is a weighted average of the difference within each stratum. Estimates from the 2 strata (tobacco user, tobacco non-user) were combined with Cochran-Mantel-Haenszel (CMH) weights

2. Secondary Outcome: Percentage of Participants Who Were Overall Responders at Week 24
Description: Overall responders were defined as participants with a ≥2 mm reduction in proptosis AND a ≥2 point reduction in Clinical Activity Score (CAS) from Baseline in the study eye, without deterioration (≥2 mm increase in proptosis or ≥2 point increase in CAS) in the fellow eye at Week 24.
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to active (inflammatory phase) thyroid eye disease/ Graves' Ophthalmopathy or Orbitopathy (TED/GO); 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active (inflammatory phase) TED/GO (ignore "equivocal" redness); 6. Chemosis; 7. Inflammation of caruncle or plica. Each item is scored (1=present; 0=absent) and scores for each item are summed for total score of 0 (no clinical activity) to 7 (most clinical activity).
Time Frame: Week 24
Population: Intent-to-treat population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Number analyzed (Participants) | 42 | 41
percentage of participants | 7.1 | 78.0
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab 20 mg/kg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Two-sided p-value calculated assuming the test statistic was distributed as a standard normal random variable; Stratified difference in percentages = 70.82, 95% CI 2-sided [55.89 to 85.75], Standard Error of Mean 7.62 — Stratified difference (teprotumumab - placebo) is a weighted average of the difference within each stratum. Estimates from the 2 strata (tobacco user, tobacco non-user) were combined with CMH weights

3. Secondary Outcome: Percentage of Participants Who Were CAS Categorical Responders at Week 24 (Study Eye)
Description: CAS categorical responders were defined as participants with a reduction to a CAS of 0 or 1 (no or minimal inflammatory symptoms) in study eye.
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to active (inflammatory phase) thyroid eye disease/ Graves' Ophthalmopathy or Orbitopathy (TED/GO); 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active (inflammatory phase) TED/GO (ignore "equivocal" redness); 6. Chemosis; 7. Inflammation of caruncle or plica. Each item is scored (1=present; 0=absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms).
Time Frame: Week 24
Population: Intent-to-treat population: all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Number analyzed (Participants) | 42 | 41
percentage of participants | 21.4 | 58.5
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab 20 mg/kg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Two-sided p-value calculated assuming the test statistic was distributed as a standard normal random variable; Stratified difference in percentages = 36.03, 95% CI 2-sided [17.39 to 54.67], Standard Error of Mean 9.51 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Proptosis to Week 24 (Study Eye)
Time Frame: Baseline, up to Week 24
Population: Intent-to-treat population: all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Number analyzed (Participants) | 42 | 41
mm | -0.54 (0.192) | -2.82 (0.191)
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab 20 mg/kg; Test type: Superiority; p < 0.001, mixed model for repeated measures (MMRM) — Results obtained from an MMRM with an unstructured covariance matrix including the following terms: Baseline value, tobacco use status, treatment group, visit, visit-by-treatment interaction and visit-by-Baseline-value interaction; LS mean difference = -2.28, 95% CI 2-sided [-2.77 to -1.80], Standard Error of Mean 0.244

5. Secondary Outcome: Percentage of Participants Who Were Diplopia Responders at Week 24
Description: Diplopia responders were defined as participants with Baseline diplopia Subjective Diplopia Score grade >0 in the study eye who had a reduction of ≥1 grade with no corresponding deterioration (≥1 grade worsening) in the fellow eye at Week 24. Denominator is the number of subjects with diplopia at Baseline.
  The Subjective Diplopia Score is a clinical measure of diplopia severity on a grade scale of 0 to 3: 0=no diplopia; 1=intermittent (diplopia in primary position of gaze, when tired or when first awakening); 2=inconstant (diplopia at extremes of gaze); 3=constant (continuous diplopia in primary or reading position).
Time Frame: Week 24
Population: Intent-to-treat population: all randomized participants with diplopia at baseline in the study eye.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Number analyzed (Participants) | 28 | 28
percentage of participants | 28.6 | 67.9
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab 20 mg/kg; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel — Two-sided p-value calculated assuming the test statistic was distributed as a standard normal random variable; Stratified difference in percentages = 39.29, 95% CI 2-sided [15.55 to 63.02], Standard Error of Mean 12.11 — Stratified difference is a weighted average of the difference within each stratum. Estimates from the 2 strata (tobacco user, tobacco non-user) were combined with CMH weights

6. Secondary Outcome: Change From Baseline in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Questionnaire Overall Score to Week 24
Description: The GO-QoL is a 16-item self-administered questionnaire divided into 2 subsets and used to assess the perceived effects of TED by the subjects on (i) their daily physical activity as it relates to visual function, and (ii) psychosocial functioning. The range of the GO-QoL overall transformed scores is 0 to 100, where higher values correspond to better quality of life.
Time Frame: Baseline, up to Week 24
Population: Intent-to-treat population: all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Teprotumumab 20 mg/kg
Number analyzed (Participants) | 42 | 41
score on a scale | 4.43 (2.102) | 13.79 (2.074)
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab 20 mg/kg; Test type: Superiority; p < 0.001, mixed model for repeated measures (MMRM) — [p-value comment as in outcome 4, analysis 1]; Difference in LS mean = 9.36, 95% CI 2-sided [4.08 to 14.64], Standard Error of Mean 2.651

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of the Double-Masked Treatment Period (up to 24 weeks) plus 3 weeks.
Arm/Group | Placebo | Teprotumumab 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/42 | 2/41
Other Adverse Events (participants affected / at risk) | 29/42 | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | Teprotumumab 20 mg/kg (N=41)
Visual field defect (Nervous system disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | Teprotumumab 20 mg/kg (N=41)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 4 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 1 | 5
Influenza (Infections and infestations) | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 14
Dizziness (Nervous system disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 4 | 4
Amenorrhoea (Reproductive system and breast disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 10
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 5
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT03298867/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT03298867/SAP_001.pdf